CLINICAL TRIAL: NCT02877953
Title: Transitional Care Interventions Post-TIPS
Brief Title: Transitional Care Interventions for Patients With Cirrhosis Post-TIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shihezi University (Other)
Responsible Party: Principal Investigator, HOU Wei-wei, Director, Shihezi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCI-2016
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The conventional care was performed for the patients of control group
- Intervention group (Experimental): the prevention of complications post-TIPS
  Interventions: Behavioral: the prevention of complications post-TIPS

INTERVENTIONS:
Behavioral: the prevention of complications post-TIPS — Continuous nursing through telephone follow-up, family visits, and WeChat guided patients to prevent gastrointestinal bleeding, infection and constipation ,intake quality low-protein diet, recognize minimal encephalopathy, monitor blood ammonia, return visit regularly, deal with adverse drug reactions of anticoagulant.
  Arms: Intervention group

SUMMARY:
The investigators conducted a randomized controlled trial to describe if multidisciplinary and patient-centered transitional care interventions for patients with cirrhosis post-TIPS can improve compliance behavior and reduce complications post-TIPS after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diagnosis of cirrhosis;
* Child-Pugh Score <10;
* Informed Consent.

Exclusion Criteria:

* Age <18 years;
* Right ventricular failure;
* Severe systemic infection;
* Hepatocellular carcinoma (HCC);
* Terminal disease; and
* Failure to provide written consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The compliance behavior associated with complications post-TIPS | 1 and 3 months after discharge
  It was surveyed using a self-designed questionnaire based on evidence. The questionnaire includes 6 items that address taking medicine on time, quality low-protein diet intake, going to sleep at a regular time, moderate exercise, emotion regulation, regular follow-up. Item responses are on a 4-point scale (0 = never to 3 = always). Data were collected by face-to-face interviews with trained transition nurses. Change is being assessed

SECONDARY OUTCOMES:
incidence of adverse events (shunt dysfunction and hepatic encephalopathy) | 1 and 3 months after discharge
  Change is being assessed
Child-Pugh scores | Baseline, 1 and 3 months after discharge
  Change is being assessed
Blood ammonia levels | Baseline, 1 and 3 months after discharge
  Change is being assessed

IPD SHARING:
Plan to Share IPD: Undecided
According to the actual situation to decide whether to share data

REFERENCES:
- [Derived] Yang R, Xu Y, Hou W, Wang L, Xiao S, Li C, Shao H, Fei X, Wang Z. Transitional Care for Patients With Portal Hypertension: A Multicenter Study of Intervention for Post-TIPS Patients. Clin Nurs Res. 2023 May;32(4):785-796. doi: 10.1177/10547738221112746. Epub 2022 Sep 1. PMID 36047431